CLINICAL TRIAL: NCT03496103
Title: Induction of Innate Neutrophilic Nasal Inflammation in a Pollen Exposure Chamber
Brief Title: Innate Neutrophilic Nasal Inflammation in a Pollen Exposure Chamber
Acronym: Pollen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: Pollen Exposure Chamber
Record Dates: First submitted 2018-04-03; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — ragweed pollen

STUDY DESIGN:
Intervention Model Description: Healthy non allergic and ragweed allergic subjects were exposed to ragweed pollen in a pollen exposure chamber for 3 hrs and symptom score was recorded
Masking Description: Investigator received de-identified biological material for further studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allergic Subjects (Other): After recording baseline symptoms, subjects were exposed to ragweed pollen for three hours and symptoms were recorded
  Interventions: Biological: ragweed pollen
- Healthy (Other): After recording baseline symptoms, subjects were exposed to ragweed pollen for three hours and symptoms were recorded
  Interventions: Biological: ragweed pollen

INTERVENTIONS:
Biological: ragweed pollen — three hours ragweed pollen in a allergen exposure chamber

SUMMARY:
In this study subjects self recorded nasal and ocular symptoms scores from exposure to ragweed pollen in an Allergen Challenge Chamber (ACC). This single site study of seasonal allergic rhinitis was designed to enroll up to 35 participants. These participants would be age 18-70, male and female, with a mixture of ethnic groups. The study would involve 2 phases: Screening and Exposure. In the Exposure phase, participants were exposed to pollen for up to 180 minutes.

DETAILED DESCRIPTION:
This was a study to evaluate self recorded nasal and ocular allergy symptom scores from exposure to ragweed pollen in an Allergen Challenge Chamber (ACC). This single site study of seasonal allergic rhinitis was designed to enroll up to 35 participants. These participants would be age 18-70, male and female, with a mixture of ethnic groups. The study would involve 2 phases: Screening and Exposure. In the Exposure phase, participants were exposed to pollen for up to 180 minutes. For allergic participants, qualification symptom scores at 120 minutes of exposure determined if ACC exposure would be continued.

ELIGIBILITY:
Inclusion Criteria:

1. Participant demonstrates understanding of the study and has provided an appropriately signed and dated informed consent.
2. Male or Female, 18 to 70 years of age, at time of the Screening visit.
3. Positive allergic participants must have a history of at least moderate AR due to hypersensitivity to ragweed pollen for a minimum of 2 years prior to the Screening visit.
4. Positive allergic participants must respond to the ragweed pollen through a standard SPT administered at the Screening visit. A positive SPT is defined as a specified aeroallergen wheal diameter of at least 5 mm or larger than the negative control (normal saline). A historical SPT performed within three-hundred sixty-five (365) days or one (1) year will be accepted in lieu of performing a new SPT.
5. Normal negative control participants must have no medical history suggestive of chronic or recurrent nasal and ocular symptoms secondary to allergy to the ragweed pollen.
6. Normal negative control participants must demonstrate a negative SPT to the ragweed pollen at the Screening visit. A historical SPT performed within three-hundred sixty-five (365) days or one (1) year will be accepted in lieu of performing a new SPT.
7. Subject understands and is willing, able and likely to comply with study procedures and restrictions.
8. Subject, if female of child bearing potential, must have a negative urine pregnancy test at Visit 1. All females of child bearing potential must agree to a medically acceptable form of birth control throughout the study duration and for at least 1 month prior to Visit 1. Acceptable methods of birth control for this study include:

   1. oral, patch, or intra-vaginal contraceptives
   2. Norplant System®
   3. Depo-Provera®
   4. Intrauterine device (IUD)
   5. double barrier method
   6. abstinence
   7. surgically sterile females (hysterectomy or tubal ligation)
   8. > 1 year post-menopausal females
   9. abstinence
9. Other than SAR, participant is healthy as determined by pre-study medical history, physical examination and vital signs. Any chronic conditions that may interfere with the study outcomes or the subject's safety will be considered clinically significant and a reason for exclusion.
10. Subject must be able to read, comprehend, and record all information in English.

Exclusion Criteria:

1. Has significant current nasal or ocular symptoms that the study doctor associates with perennial allergic or non-allergic rhinitis.
2. Female participant who is pregnant or lactating.
3. Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study. This includes a clinically relevant medical or surgical history or presence of other respiratory disease (exceptions made for asthma and AR as defined in further exclusion criteria), or gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, immunological, dermatological, connective tissue diseases or disorders, or a history of malignancy within the past 5 years, with the exception of non- melanoma skin cancer.
4. Has any significant abnormalities found during physical exam as determined by the investigator.
5. Has had a respiratory and/or bacterial sinusitis infection during the past one (1) week prior to the first challenge visit or any subsequent study visits.
6. Has a current medical history of significant pulmonary disease and/or active asthma requiring daily drug therapy. Mild, intermittent asthma is permitted (managed with short acting beta-agonist less than 3 times per week). Isolated exercise-induced bronchospasm is also permitted.
7. Has received an investigational drug within the last thirty (30) days.
8. Has a history of rebound nasal congestion from extended use of topical decongestants.
9. Has had use of immunotherapy containing short ragweed within the last 3 years.
10. Has a history of nasal polyps, nasal septal perforation, or nasal tract malformations as noted on physical exam.
11. Has a clinically significant history of substance abuse, drug addiction, or alcohol abuse in the past 3 years in the judgement of the investigator.
12. Currently uses or is expected to use any of the disallowed medications as listed in Disallowed Medications in section 4.3.
13. Cannot communicate reliably with the investigator.
14. Is unlikely to cooperate with the requirements of the study.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2016-03-12 (Actual); Study Completion 2016-03-12 (Actual)

PRIMARY OUTCOMES:
Effect of ragweed pollen exposure | 3 hours
  Subjects self-recorded nasal allergy symptom scores from exposure to ragweed pollen in an Allergen Challenge Chamber (ACC). The subjects self-assessed total nasal symptom scores, a combination or runny nose, itchy nose, sneezing and nasal congestion on a scale of 0-3 using the Likert 4-point severity score: 0=none, 1=minimal, 2=moderate, 3=severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Sur, MD, Principal Investigator — University of Texas